CLINICAL TRIAL: NCT01844388
Title: A Study to Compare a New Eye Drop Formulation With Refresh Contacts®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10077X-001
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Contact Lens Lubrication

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carboxymethylcellulose Based Eye Drop Formula (Experimental): 1-2 drops of carboxymethylcellulose based eye drop formula in each eye, a minimum of 4 times a day for 90 days. One of the 4 times a day may be to prepare the contact lens for insertion.
  Interventions: Drug: carboxymethylcellulose based eye drop formula
- REFRESH CONTACTS® (Active Comparator): 1-2 drops carboxymethylcellulose sodium based eye drop solution (REFRESH CONTACTS®) in each eye, a minimum of 4 times a day for 90 days. One of the 4 times a day may be to prepare the contact lens for insertion.
  Interventions: Drug: carboxymethylcellulose sodium based eye drop solution

INTERVENTIONS:
Drug: carboxymethylcellulose based eye drop formula — 1-2 drops of carboxymethylcellulose based eye drop formula in each eye, a minimum of 4 times a day for 90 days. One of the 4 times a day may be to prepare the contact lens for insertion.
  Arms: Carboxymethylcellulose Based Eye Drop Formula
Drug: carboxymethylcellulose sodium based eye drop solution — 1-2 drops carboxymethylcellulose sodium based eye drop solution (REFRESH CONTACTS®) in each eye, a minimum of 4 times a day for 90 days. One of the 4 times a day may be to prepare the contact lens for insertion.
  Other Names: REFRESH CONTACTS®
  Arms: REFRESH CONTACTS®

SUMMARY:
This study will compare the safety and efficacy of a new carboxymethylcellulose based eye drop formula to Refresh Contacts® for lubricating and rewetting contact lenses.

ELIGIBILITY:
Inclusion Criteria:

-Adapted contact wearer with daily usage of at least 6 hours a day, 5 days a week.

Exclusion Criteria:

* Wearing monovision lenses
* Have had refractive surgery within the previous 12 months
* Have infection of the eye, eyelids or eye structures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2013-05-29 (Actual); Primary Completion 2013-12-02 (Actual); Study Completion 2013-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Bloomington, Illinois, United States

REFERENCES:
- [Background] Nichols JJ, Lievens CW, Bloomenstein MR, Liu H, Simmons P, Vehige J. Dual-Polymer Drops, Contact Lens Comfort, and Lid Wiper Epitheliopathy. Optom Vis Sci. 2016 Aug;93(8):979-86. doi: 10.1097/OPX.0000000000000878. PMID 27254807

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carboxymethylcellulose Based Eye Drop Formula | REFRESH CONTACTS®
Started | 244 | 121
Completed | 236 | 114
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboxymethylcellulose Based Eye Drop Formula | REFRESH CONTACTS® | Total
Number analyzed (Participants) | 244 | 121 | 365
Age, Customized [Number; unit: participants]
  <40 years | 170 | 90 | 260
  ≥40 years | 74 | 31 | 105
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 90 | 272
  Male | 62 | 31 | 93

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Contact Lens Distance Visual Acuity Change From Baseline
Description: Contact lens distance visual acuity was measured for each eye using the LogMAR visual acuity eye chart. The worse eye at Baseline was used for analysis. A change of 0.1 on the LogMAR scale was equivalent to a 1 line change in visual acuity. The following categories are reported: Better=an increase in 2 or more lines, No Change=a change of +/- 1 line, and Worse=a decrease of 2 lines or more.
Time Frame: Baseline, Day 90
Population: Intent-to-treat Population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Carboxymethylcellulose Based Eye Drop Formula | REFRESH CONTACTS®
Number analyzed (Participants) | 244 | 121
percentage of participants
  Better | 11.1 | 10.7
  No Change | 88.9 | 88.4
  Worse | 0.0 | 0.8

2. Other Pre Specified Outcome: Average Daily Contact Wearing Time
Description: The average reported number of hours per day that contact lenses were worn by participants during the previous 7 days.
Time Frame: Day 90
Population: Completed population included all enrolled participants who received study treatment and completed the study through Day 90.
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Carboxymethylcellulose Based Eye Drop Formula | REFRESH CONTACTS®
Number analyzed (Participants) | 236 | 114
hours per day | 13.8 (2.59) | 13.9 (3.01)

3. Other Pre Specified Outcome: Reason for Contact Lens Replacement
Description: The reason the contact lens needed to be replaced was recorded for each eye. The following categories are reported: Scheduled Replacement, Discomfort, Lens Damage, Unacceptable Vision and Lens Lost. There may be multiple reasons for replacement of the contact lens for a single eye.
Time Frame: Day 90
Population: as for outcome 2
Measure: Number; unit: eyes
Units Other Than Participants: Contact Lenses Replaced
Arm/Group | Carboxymethylcellulose Based Eye Drop Formula | REFRESH CONTACTS®
Number analyzed (Participants) | 236 | 114
Number analyzed (Contact Lenses Replaced) | 177 | 86
eyes
  Scheduled Replacement | 158 | 74
  Discomfort | 11 | 5
  Lens Damage | 9 | 7
  Unacceptable Vision | 1 | 0
  Lens Lost | 4 | 0

ADVERSE EVENTS:
Description: Treatment-emergent adverse events (adverse events which occur after study drug is first administered) are reported.
Arm/Group | Carboxymethylcellulose Based Eye Drop Formula | REFRESH CONTACTS®
Serious Adverse Events (participants affected / at risk) | 1/244 | 0/121
Other Adverse Events (participants affected / at risk) | 0/244 | 0/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Carboxymethylcellulose Based Eye Drop Formula (N=244) | REFRESH CONTACTS® (N=121)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/182 | 0/90 — Not treatment-related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.